CLINICAL TRIAL: NCT05111184
Title: Educational Impact of a Tablet Application on Nutrition in Maintenance Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Waid City Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WaidCH
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internvention group (Other)
  Interventions: Behavioral: Education groupe

INTERVENTIONS:
Behavioral: Education groupe — Education

SUMMARY:
The investigator examines of the impact of digital training on the sodium, potassium and phosphate content of various foods in dialysis patients. The training takes place visually as self-study in the form of a computer-based application.

The working hypothesis is that trained dialysis patients have consistently better plasma electrolyte values than untrained participants.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis Patient

Exclusion Criteria:

* Pregnancy
* Not preparing own meals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change of electrolyte levels | one month